CLINICAL TRIAL: NCT03445546
Title: Platelet Function in Resuscitated Patients-2
Status: Completed | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: 28-291 ex15/16
Record Dates: First submitted 2018-02-16; First posted 2018-02-26 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Acute Myocardial Infarction; Cardiac Arrest
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- oral P2Y12 inhibition: Patients with cardiac arrest and myocardial infarction treated with oral P2Y12 Inhibitor (from the historic cohort of NCT02914795)
  Interventions: Diagnostic Test: diagnostic test of platelet function
- intravenous P2Y12 inhibition: Patients with cardiac arrest and myocardial infarction treated with intravenous P2Y12 Inhibitor (cangrelor)
  Interventions: Diagnostic Test: diagnostic test of platelet function

INTERVENTIONS:
Diagnostic Test: diagnostic test of platelet function — Light transmittance aggregometry and VerifyNow

SUMMARY:
Approx. 65% of resuscitated patients at the intensive care unit for internal medicine are due to myocardial infarction. Almost all patients are initially diagnosed and treated in the cath lab. Therapy usually consists of one or more stent implantations. After implantation of a coronary stent, dual platelet inhibition is necessary for 12 months. Insufficient platelet inhibition causes an pronounced increase in risk of stent thrombosis. Therefore, secured inhibition and knowledge of the individual platelet function is valuable.

DETAILED DESCRIPTION:
Patients after successful resuscitation associated to a myocardial infarction will be included into the study the morning after the index event. Patients get dual platelet inhibition using cangrelor as P2Y12 (purinergic G protein-coupled receptors-12) inhibitor plus acetylsalicylic acid (ASS). Patients are treated with therapeutic hypothermia according to the local Standard operating procedure for 24h and rewarming is performed within an additional 5 to 20h. Platelet function is measured every morning and ASS mediated as well as P2Y12 mediated platelet function inhibition is recorded. All relevant clinical data including APACHE (Acute Physiology and Chronic Health Evaluation) and SOFA (Sequential Organ Failure Assessment score) scores are collected.

The degree of platelet inhibition over time (4 days) and differences between the three drugs tested will be evaluated by optical aggregometry and by using the commercial VerifyNow test system.

ELIGIBILITY:
Inclusion Criteria:

* Myocardial infarction
* dual platelet inhibition
* resuscitation
* therapeutic hypothermia

Exclusion Criteria:

* none

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients surviving the first night after resuscitation due to myocardial infarction
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2018-05-15 (Actual); Study Completion 2018-05-15 (Actual)

PRIMARY OUTCOMES:
Platelet inhibition measured with optical aggregometry | 4 days
  Light transmittance aggregometry

SECONDARY OUTCOMES:
Composite of death and stent thrombosis | 4 days
  Composite of death and stent thrombosis

CONTACTS AND LOCATIONS:
Overall Officials: Dirk von Lewinski, MD, Principal Investigator — Medical University of Graz
Locations (1):
- Medical University of Graz, Graz, Austria

REFERENCES:
- [Result] Bhatt DL, Lincoff AM, Gibson CM, Stone GW, McNulty S, Montalescot G, Kleiman NS, Goodman SG, White HD, Mahaffey KW, Pollack CV Jr, Manoukian SV, Widimsky P, Chew DP, Cura F, Manukov I, Tousek F, Jafar MZ, Arneja J, Skerjanec S, Harrington RA; CHAMPION PLATFORM Investigators. Intravenous platelet blockade with cangrelor during PCI. N Engl J Med. 2009 Dec 10;361(24):2330-41. doi: 10.1056/NEJMoa0908629. PMID 19915222
- [Result] Angiolillo DJ, Schneider DJ, Bhatt DL, French WJ, Price MJ, Saucedo JF, Shaburishvili T, Huber K, Prats J, Liu T, Harrington RA, Becker RC. Pharmacodynamic effects of cangrelor and clopidogrel: the platelet function substudy from the cangrelor versus standard therapy to achieve optimal management of platelet inhibition (CHAMPION) trials. J Thromb Thrombolysis. 2012 Jul;34(1):44-55. doi: 10.1007/s11239-012-0737-3. PMID 22569899
- [Result] White HD, Bhatt DL, Gibson CM, Hamm CW, Mahaffey KW, Price MJ, Steg PG, Stone GW, Cortese B, Wilensky M, Deliargyris EN, Liu T, Prats J, Harrington RA. Outcomes with cangrelor versus clopidogrel on a background of bivalirudin: insights from the CHAMPION PHOENIX (A Clinical Trial Comparing Cangrelor to Clopidogrel Standard Therapy in Subjects Who Require Percutaneous Coronary Intervention [PCI]). JACC Cardiovasc Interv. 2015 Mar;8(3):424-433. doi: 10.1016/j.jcin.2014.09.025. Epub 2015 Feb 18. PMID 25703887
- [Result] Nolan JP, Soar J, Cariou A, Cronberg T, Moulaert VR, Deakin CD, Bottiger BW, Friberg H, Sunde K, Sandroni C. European Resuscitation Council and European Society of Intensive Care Medicine Guidelines for Post-resuscitation Care 2015: Section 5 of the European Resuscitation Council Guidelines for Resuscitation 2015. Resuscitation. 2015 Oct;95:202-22. doi: 10.1016/j.resuscitation.2015.07.018. No abstract available. PMID 26477702
- [Result] Roffi M, Patrono C, Collet JP, Mueller C, Valgimigli M, Andreotti F, Bax JJ, Borger MA, Brotons C, Chew DP, Gencer B, Hasenfuss G, Kjeldsen K, Lancellotti P, Landmesser U, Mehilli J, Mukherjee D, Storey RF, Windecker S; ESC Scientific Document Group. 2015 ESC Guidelines for the management of acute coronary syndromes in patients presenting without persistent ST-segment elevation: Task Force for the Management of Acute Coronary Syndromes in Patients Presenting without Persistent ST-Segment Elevation of the European Society of Cardiology (ESC). Eur Heart J. 2016 Jan 14;37(3):267-315. doi: 10.1093/eurheartj/ehv320. Epub 2015 Aug 29. No abstract available. PMID 26320110
- [Result] Nikolaou NI, Arntz HR, Bellou A, Beygui F, Bossaert LL, Cariou A; Initial management of acute coronary syndromes section Collaborator. European Resuscitation Council Guidelines for Resuscitation 2015 Section 8. Initial management of acute coronary syndromes. Resuscitation. 2015 Oct;95:264-77. doi: 10.1016/j.resuscitation.2015.07.030. Epub 2015 Oct 15. No abstract available. PMID 26477416
- [Result] Task Force on the management of ST-segment elevation acute myocardial infarction of the European Society of Cardiology (ESC); Steg PG, James SK, Atar D, Badano LP, Blomstrom-Lundqvist C, Borger MA, Di Mario C, Dickstein K, Ducrocq G, Fernandez-Aviles F, Gershlick AH, Giannuzzi P, Halvorsen S, Huber K, Juni P, Kastrati A, Knuuti J, Lenzen MJ, Mahaffey KW, Valgimigli M, van 't Hof A, Widimsky P, Zahger D. ESC Guidelines for the management of acute myocardial infarction in patients presenting with ST-segment elevation. Eur Heart J. 2012 Oct;33(20):2569-619. doi: 10.1093/eurheartj/ehs215. Epub 2012 Aug 24. No abstract available. PMID 22922416
- [Derived] Pruller F, Bis L, Milke OL, Fruhwald F, Patzold S, Altmanninger-Sock S, Siller-Matula J, von Lewinski F, Ablasser K, Sacherer M, von Lewinski D. Cangrelor Induces More Potent Platelet Inhibition without Increasing Bleeding in Resuscitated Patients. J Clin Med. 2018 Nov 15;7(11):442. doi: 10.3390/jcm7110442. PMID 30445678